CLINICAL TRIAL: NCT05553561
Title: Therapeutic Effect of Intense Regulated Pulse Light in Patients With Dry Eye Disease
Brief Title: Intense Regulated Pulse Light Therapy in Dry Eye Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Rofaida Mostafa Mansour Serag EL Deen, Ophthalmologist at Menoufia university hospitals, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7/2022OPHT23
Record Dates: First submitted 2022-09-07; First posted 2022-09-23 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Dry Eye Disease
Keywords: IPL therapy; IRPL therapy; Dry eye; MGD
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IRPL Therapy (Active Comparator): 17 patients with moderate to severe evaporative dry eye disease will treated with 3 sessions of IRPL therapy.
  Interventions: Procedure: IPRL device
- Non IRPL Therapy (Active Comparator): 17 patients with moderate to severe evaporative dry eye disease will treated with traditional methods of MGD
  Interventions: Procedure: pharmacological therapy & Eyelid hygiene

INTERVENTIONS:
Procedure: IPRL device — Intense pulsed light therapy (IPL) is a non-coherent large wavelength high-intensity light in the range of 500-1200nm. It has been used by many investigators for the treatment of evaporative dry eye safely and effectively.
  Arms: IRPL Therapy
Procedure: pharmacological therapy & Eyelid hygiene — traditional methods of MGD treatment as Eyelid hygiene, topical preservative free lubricant, topical & systemic antibiotics & anti-inflammatory agent
  Arms: Non IRPL Therapy

SUMMARY:
The aim of this study is to assess the effect of intense regulated pulse light (IRPL) on the treatment of Dry eye.

DETAILED DESCRIPTION:
Dry eye disease is a common ocular condition that needs prompt diagnosis and careful treatment interventions. If left untreated, it can lead to numerous sight threatening complications, including ulceration of the cornea, blepharitis, alterations of the tear film, conjunctivitis, and in severe cases, significant drying of the eye may lead to scarring, thinning, and even perforation of the cornea.

Intense pulsed light (IPL) therapy is a new treatment strategy for treatment of MGD by inducing the restoration of the normal activity of the meibomian glands. In fact, IPL has been used for treating the patients with facial telangiectasias and erythema of rosacea and also resulted in improvement in ocular surface health.

Evaporative form is the commonest form of DED and it is mainly caused by meibomian glands dysfunction (MGD). The usual traditional treatment options for MGD include warm compresses, expression of meibomian glands (MG), anti-inflammatory drugs, and lubricant eye drops.

The aim of this study is to assess the effect of intense regulated pulse light (IRPL) on the treatment of Dry eye.

The study included 34 patients with moderate to severe evaporative dry eye. The symptoms will be assessed with the Dry Eye-Related Quality of Life Score (DEQ-5) Questionnaire. The tear film will be assessed through MediWorks D130+S390L (WDR) which is a device attached to the slit lamp for non-invasive examination of tear film.

Patients will be divided into 2 groups: The 1st group include (17) patients who will be treated with Intense Regulated Pulse Light (IRPL) & the 2nd group include (17) patients will treated by traditional methods of MGD as Eyelid hygiene, topical lubricant, topical & systemic antibiotics & anti-inflammatory agents

IRPL will be done using E-Eye (E-Swin, France) & each patient will undergo 3 sessions on Day (1), Day (15), and Day (45).

The patients will be reassessed after the 3rd session.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe dry eye disease & clinicaily significant signs of meibomian gland dysfunction

Exclusion Criteria:

* Use systemic medications known to affect the eye two weeks prior to baseline assessment.
* Pregnancy.
* Ocular surgery or dermatologic treatments in the previous Two months or during the treatment period.
* Implants, tattoos, or pigmented lesions in the treatment area.
* Contraindications to IPL therapy, including the use of photosensitive medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Non-invasive tear film break up time | before treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Change in Non-invasive tear film break up time | Within 1 month after completion of treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Tear Meniscus Height | before treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Change in Tear Meniscus Height | Within 1 month after completion of treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Lipid layer thickness | before treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Change in Lipid layer thickness | Within 1 month after completion of treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Meibomian glands % loss grading | before treatment
  assessment of tear film through MediWorks device attached to the slitlamp
Change in Meibomian glands % loss grading | Within 1 month after completion of treatment
  assessment of tear film through MediWorks device attached to the slitlamp
patient's quality of life affection | before treatment
  The effect of dry eye on the patient's Quality Of Life was evaluated with the aid of Dry Eye-Related Quality of Life Score (DEQ-5) Questionnaire.
Change in patient's quality of life affection | Within 1 month after completion of treatment
  The effect of dry eye on the patient's Quality Of Life was evaluated with the aid of Dry Eye-Related Quality of Life Score (DEQ-5) Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Monoufia university, Menoufia, Egypt